CLINICAL TRIAL: NCT01158950
Title: A Randomized, Double-Blind Study of Neural Circuit Responses to COMT Inhibitors
Brief Title: A Study of Neural Circuit Responses to Catechol-O-methyl Transferase (COMT) Inhibitors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Berkeley (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2009-12-461; W81XWH-10-1-0231 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2010-07-07; First posted 2010-07-08 (Estimated); Results first posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Impulsive Behavior
MeSH Terms: conditions — Impulsive Behavior | interventions — Tolcapone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tolcapone (Experimental): Drug: Tolcapone 200mg (single dose) administered at study visit
  Interventions: Drug: Tolcapone
- Placebo (Placebo Comparator): Drug: Placebo for tolcapone administered at study visit
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tolcapone — Drug: Tolcapone 200mg (single dose) administered at study visit
  Other Names: Tasmar
  Arms: Tolcapone
Other: Placebo — Placebo (200mg) administered at study visit
  Arms: Placebo

SUMMARY:
In this study, we seek to understand the effects of tolcapone, an FDA-approved COMT inhibitor, on reward choice and response inhibition, two measures we have previously shown to be altered in subjects with alcoholism. We now plan to test the hypothesis that COMT regulation of cortical dopamine levels is critical for regulation financial choices. Specifically, we propose that the lower levels of cortical dopamine present in individuals with the val158val COMT genotype reduces the inhibitory effect of frontal cortical areas on impulsive choice; an idea that extends previous hypotheses about the negative consequences of decreased prefrontal dopamine levels on inhibitory control. Moreover, this hypothesis suggests that inhibiting COMT may slow the degradation of dopamine and thereby decrease impulsivity.

DETAILED DESCRIPTION:
Drug consumption despite adverse consequences is a defining feature of human addiction (DSM-IV-TR, 2004). Impulsivity, a tendency to choose an immediate action despite delayed adverse consequences, is a major risk factor for tobacco, psychostimulant, opioid and alcohol abuse. In humans, impulsivity can be quantified by presenting subjects with a choice between a small immediate monetary reward or a larger but delayed reward. We recently found that the val158val allele for the enzyme catechol-O-methyltransferase (COMT), which is associated with more rapid cortical dopamine catabolism and thus lower cortical dopamine levels correlates with greater impulsivity and greater fMRI blood oxygen level dependent (BOLD) signal in dorsolateral prefrontal and posterior parietal cortices.

The first phase of the study will involve healthy controls. The second phase of the study will involve abstinent alcoholics matched for age, education, and gender. Subjects will range in age between 18 and 50 years old.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years.
* Subject is right-handed.
* If female, subject is non-lactating, not pregnant, and using a reliable contraception method (i.e. abstinence, intrauterine device (IUD), hormonal birth control or barrier method).
* Subject is able to read and speak English.
* Subject is a high school graduate.
* Subject is able and willing to provide written and informed consent.
* Subject is able to understand and follow the instructions of the investigator, and understand all ratings scales.
* Subject is in good health.

Exclusion Criteria:

* Using cocaine, stimulants (other than THC, nicotine, & caffeine)amphetamines, hallucinogens, "ecstasy", opiates, sedatives, pain pills, sleeping pills or other psychoactive drugs within two weeks of the start of the study OR more than 10 times in the last year.
* Has a current dependence on, or addiction to any psychoactive drug (except nicotine or caffeine) including alcohol.
* Clinically significant medical or psychiatric illness requiring treatment as determined by screening blood tests, medical history, and physical exam performed or reviewed by the study physician.
* Subject has a history of major alcohol related complications within the proceeding 2 years (liver failure/cirrhosis, pancreatitis, esophageal varices, etc.)
* Liver function test ≥ 3 times normal upper limit.
* BAC level > 0.05% at the beginning of screening visit (within margin of error of detection).
* Has a neurological dysfunction or psychiatric disorder.
* Has severe low blood pressure.
* Has uncontrolled high blood pressure.
* Regular use of any of the drugs on the tolcapone or entacapone contraindications list OR within 2 weeks of drug administration.
* Regular use of SSRIs.
* Has an allergy or intolerance to tolcapone or entacapone.
* Subject has received an investigational drug within 30 days of screening visit.
* Subject is considered unsuitable for the study in the opinion of the investigator or study physician for any other reason.

MRI Exclusion Criteria:

* The subject has metal (metal plates, pins, wires or screws, artificial limb, joint replacement or anything that might have been inserted during an operation) in his/her body.
* Subject has a pacemaker, defibrillator, stent, or any metal implants related to heart/blood flow problems.
* Subject has worked with metals (ie. metallurgy, metal shaving, welding, soldering, etc).
* Subject has been wounded with anything metal (bullet, shrapnel or metal filling).
* Has ever gotten a piece of metal in the eye.
* Has tattoos done with ink containing metal or permanent eyeliner.
* Wears color contact lenses.
* Has a hearing problem or hearing aid, cochlear implant or past ear surgery.
* Has any irremovable dental bridges, dental plates, metal caps or any other non-removable metal in the mouth.
* The subject is claustrophobic.
* The subject is pregnant. (women only)
* Has a IUD. (women only)
* Significantly overweight.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Fields, MD, PhD, Principal Investigator — UCSF: Ernest Gallo Clinic and Research Center; Jennifer Mitchell, PhD, Study Director — UCSF: Ernest Gallo Clinic and Research
Locations (2):
- United States (2):
  - University of California, Berkeley, Berkeley, California
  - UCSF: Ernest Gallo Clinic and Research Center, Emeryville, California

REFERENCES:
- [Result] Kayser AS, Allen DC, Navarro-Cebrian A, Mitchell JM, Fields HL. Dopamine, corticostriatal connectivity, and intertemporal choice. J Neurosci. 2012 Jul 4;32(27):9402-9. doi: 10.1523/JNEUROSCI.1180-12.2012. PMID 22764248

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were screened for inclusion / exclusion criteria.
Groups:
- Tolcapone First, Then Placebo: Tolcapone 200mg (single dose) then Placebo (single dose) administered at study visit, followed by crossover to other drug at next visit
- Placebo First, Then Tolcapone: Placebo (single dose) then Tolcapone 200mg (single dose) tadministered at study visit, followed by crossover to other drug at next visit
Period: 1st Intervention (1 Day)
Arm/Group | Tolcapone First, Then Placebo | Placebo First, Then Tolcapone
Started | 13 | 13
Data Collected | 12 | 11
Completed (Data included in analysis) | 12 | 11
Not Completed | 1 | 2
Not completed — Physician Decision | 1 | 2
Period: Washout (1 Week)
Arm/Group | Tolcapone First, Then Placebo | Placebo First, Then Tolcapone
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0
Period: 2nd Intervention (1 Day)
Arm/Group | Tolcapone First, Then Placebo | Placebo First, Then Tolcapone
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants receiving either Tolcapone 200mg (single dose) or Placebo (single dose) administered at study visit, followed by crossover to other drug at next visit - all participants were randomized to receive all interventions.
Arm/Group | All Study Participants
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.1 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 20
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 23
Barratt Impulsiveness Scale [Mean (Standard Deviation); unit: units on a scale] — The Barratt Impulsiveness Scale measures impulsive behavior on a 20-80 point scale, with higher numbers corresponding to greater impulsivity.
  units on a scale | 58.6 (9.1)

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between the Impulsive Choice Ratio and Baseline Impulsivity, as Measured With the Barratt Impulsiveness Scale
Description: The presented value represents a correlation. Subjects completed a delay discounting task while functional MRI images were obtained. In this task, subjects made hypothetical choices between a smaller amount of money available sooner, and a larger amount of money available later. Performance on the delay discounting task, as assessed by the impulsive choice ratio, was determined for both the tolcapone and placebo sessions, and the difference between them (tolcapone minus placebo) was calculated. This difference value was then correlated with baseline scores on the Barratt Impulsiveness Scale.
Time Frame: 120 minutes after drug ingestion
Population: The outcome for this study was the correlation between the baseline BIS score and the difference in ICR (tolcapone minus placebo). As such, one Arm/Group is presented below.
Measure: Number; unit: Correlation coefficient
Groups:
- Functional MRI Arm (Tolcapone and Placebo): This cognitive science study consists of a single arm in which all subjects receive both tolcapone and placebo in randomized, double-blind, counterbalanced, crossover fashion. Tolcapone is a medication in the class of catechol-O-methyltransferase (COMT) inhibitors. A placebo is a tablet or capsule that looks like the study medication (in this case, tolcapone) but does not contain any active ingredients.
Arm/Group | Functional MRI Arm (Tolcapone and Placebo)
Number analyzed (Participants) | 23
Correlation coefficient | -0.45
Statistical Analysis 1: Comparison: Functional MRI Arm (Tolcapone and Placebo); The comparison group represents the difference in ICR and the baseline impulsiveness scale; Test type: Superiority; p = 0.032, Fisher transformation — The threshold for statistical significance was set to p < 0.05

2. Other Pre Specified Outcome: Correlation Between the Difference in ICR (Tolcapone Minus Placebo) and the Difference in Blood Oxygen Level Dependent (BOLD) Signal in the Brain (Tolcapone Minus Placebo)
Description: The presented value represents a correlation. The difference in performance on the delay discounting task was calculated as the change in ICR (tolcapone minus placebo). In addition, the difference in BOLD activity throughout the brain was determined (tolcapone minus placebo).
Time Frame: 120 minutes after drug ingestion
Population: The outcome for this study was the correlation between the difference in the ICR and the difference in BOLD activity (tolcapone minus placebo). As such, one Arm / Group is presented below.
Measure: Number; unit: Correlation coefficient
Arm/Group | Functional MRI Arm (Tolcapone and Placebo)
Number analyzed (Participants) | 23
Correlation coefficient | -0.50
Statistical Analysis 1: Comparison: Functional MRI Arm (Tolcapone and Placebo); Test type: Superiority; p < 0.05, Fisher transformation — The threshold is set to p < 0.05, corrected for multiple comparisons; Statistical tests are computed across multiple subregions (voxels) within each area. Thus, the correlation coefficient above is a summary score

ADVERSE EVENTS:
Time Frame: 4 weeks
Groups:
- Tolcapone: Tolcapone 200mg (single dose)
- Placebo: Placebo (single dose)
Arm/Group | Tolcapone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

LIMITATIONS AND CAVEATS:
Funding constrained the number of participants. Describing the thousands of statistical tests in neuroimaging studies is not possible within this reduced format. Please see the open access pdf of Kayser et al, JNeurocience 2012.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-07-04): https://cdn.clinicaltrials.gov/large-docs/50/NCT01158950/Prot_SAP_000.pdf